CLINICAL TRIAL: NCT06427499
Title: The Clinical Investigation of Stannous Fluoride Toothpaste and a Newly Designed Toothbrush Compared to Colgate Cavity Protection Toothpaste and a Regular Toothbrush in Reducing Plaque and Gingivitis: A Three-Month Study in Thailand
Brief Title: The Clinical of Stannous Fluoride Toothpaste and a Newly Designed Toothbrush Compared to Colgate Cavity Protection Toothpaste and a Regular Toothbrush in Reducing Plaque and Gingivitis.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-04-PGN-BKS-YPZ
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Plaque; Gingivitis
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stannous Fluoride Toothpaste (Experimental)
  Interventions: Drug: Stannous fluoride toothpaste
- Colgate Cavity Protection Toothpaste (Active Comparator): MFP Fluoride toothpaste
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Stannous fluoride toothpaste — brush 2 min morning & night daily
  Arms: Stannous Fluoride Toothpaste
Drug: Colgate Cavity Protection Toothpaste — brush 2 min morning & night daily
  Arms: Colgate Cavity Protection Toothpaste

SUMMARY:
Qualified subjects will be enrolled and randomly assigned to either of the two study groups based on their initial Plaque and Gingivitis scores. During the first visit, subjects will undergo three key procedures: 1) evaluation for baseline plaque and gingivitis, 2) brushing with the assigned regimen products for two minutes, and 3) assessment for post-brushing plaque only. Subjects will be provided with clear instructions for regimen product usage and will be expected to adhere to these instructions. Follow-up evaluations for plaque and gingivitis will be conducted at one week, six weeks, and three months after initiation of regimen product use. Throughout the study period, continuous monitoring for adverse events will be carried out for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the three-month duration of the clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars). 5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
* Signed Informed Consent Form

Exclusion Criteria:

* Presence of orthodontic bands.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Pregnant or lactating subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Loe and Silness Gingival Index. | baseline, one week, six weeks and three months
  A Loe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scoreable surface and dividing that number by the total number of surfaces scored.
Quigley and Hein Plaque Index | baseline, one week, six weeks and three months
  A Quigley-Hein Plaque Index score of 0 to 5 will be assigned to all scoreable disclosed surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth score for each subject will be determined by adding the values given by the dental examiner to each scoreable surface and dividing that number by the total number of surfaces scored.

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triratana, Principal Investigator — M U International Oral Science Research, Ltd

IPD SHARING:
Plan to Share IPD: No